CLINICAL TRIAL: NCT03483103
Title: A Phase 2 Study of Lisocabtagene Maraleucel (JCAR017) as Second-Line Therapy in Adult Patients With Aggressive B-cell NHL (017006)
Brief Title: Lisocabtagene Maraleucel (JCAR017) as Second-Line Therapy (TRANSCEND-PILOT-017006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017006
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Results first posted 2022-12-29 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Nonhodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse
Keywords: JCAR017; lisocabtagene maraleucel; NHL; chimeric antigen receptor; CAR; CAR T cell; autologous T cell therapy; immunotherapy; cell therapy; liso-cel
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Lisocabtagene maraleucel at a dose of 100×10^6 CAR+ T cells (50×10^6 CD8+ CAR+ T cells and 50×10^6 CD4+ CAR+ T cells), will be given IV in a single-dose schedule on Day 1 (between 2 and 7 days following the completion of lymphodepleting chemotherapy).
  Interventions: Biological: lisocabtagene maraleucel

INTERVENTIONS:
Biological: lisocabtagene maraleucel — lisocabtagene maraleucel will be administered as a single dose intravenous (IV) injection
  Other Names: JCAR017; liso-cel

SUMMARY:
This is a Phase 2, open-label, multicenter study to determine the efficacy and safety of lisocabtagene maraleucel (JCAR017) in adult subjects who have relapsed from, or are refractory to, a single line of immunochemotherapy for aggressive B-cell non-Hodgkin lymphoma (NHL) and are ineligible for hematopoietic stem cell transplant (based on age, performance status, and/or comorbidities). Subjects will receive treatment with lisocabtagene maraleucel and will be followed for 2 years for safety, pharmacokinetics and biomarkers, disease status, quality of life, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of relapsed or refractory aggressive B-cell non-Hodgkin lymphoma of the following histology at relapse: diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS; de novo or transformed follicular lymphoma [tFL]), high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (double/triple hit lymphoma [DHL/THL]), and follicular lymphoma Grade 3B per WHO 2016 classification
* Previous treatment must include treatment with a single line of chemoimmunotherapy containing an anthracycline and a CD20-targeted agent
* Subjects must be deemed ineligible for both high-dose chemotherapy and hematopoietic stem cell transplant (based on age, performance status and/or comorbidities) while also having adequate organ function for CAR T cell treatment.
* Positron emission tomography (PET)-positive disease
* Histological confirmation of diagnosis at last relapse. Enough tumor material must be available for central confirmation of diagnosis, otherwise a new tumor biopsy is mandated.
* ECOG performance status of 0, or 1, or 2
* Adequate vascular access for leukapheresis procedure (either peripheral line or surgically-placed line)
* Subjects must agree to use appropriate contraception
* Subjects must agree to not donate blood, organs, semen, and egg cells for usage in other individuals for at least 1 year following lymphodepleting chemotherapy

Exclusion Criteria:

* Subjects with central nervous system (CNS)-only involvement by malignancy (note: subjects with secondary CNS involvement are allowed on study)
* History of another primary malignancy that has not been in remission for at least 2 years.
* Previous treatment with CD19-targeted therapy, with the exception of prior lisocabtagene maraleucel treatment in this protocol for subjects receiving retreatment
* Active hepatitis B or hepatitis C infection at the time of screening
* History of or active human immunodeficiency virus (HIV) infection at the time of screening
* Uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment at the time of leukapheresis or lisocabtagene maraleucel administration
* History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
* History or presence of clinically relevant CNS pathology
* Pregnant or nursing women
* Subject does not meet protocol-specified washout periods for prior treatments
* Prior hematopoietic stem cell transplant
* Progressive vascular tumor invasion, thrombosis, or embolism
* Venous thrombosis or embolism not managed on stable regimen of anticoagulation
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (59):
- United States (59):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Local Institution - 0043, Gilbert, Arizona
  - Scripps Clinic, La Jolla, California
  - UNC School of Medicine, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Sutter Hematology and Oncology, Sacramento, California
  - Sutter Medical Center, Sacramento, California
  - Stanford Cancer Genetics Clinic, Stanford, California
  - Local Institution - 0092, Stanford, California
  - Stanford Cancer Center, Stanford, California
  - Local Institution - 0019, Atlanta, Georgia
  - The Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - UNC School of Medicine, Atlanta, Georgia
  - Local Institution - 0003, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Local Institution - 0016, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Local Institution - 0046, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Local Institution - 0064, Louisville, Kentucky
  - Norton Cancer Institute - Brownsboro, Louisville, Kentucky
  - UNC School of Medicine, Louisville, Kentucky
  - Johns Hopkins Oncology Center Bunting Blaustein Building, Baltimore, Maryland
  - Local Institution - 0009, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Local Institution - 0052, East Brunswick, New Jersey
  - Regional Cancer Care Associates, East Brunswick, New Jersey
  - UNC School of Medicine, East Brunswick, New Jersey
  - New York Oncology Hematology - Albany Cancer Center, Albany, New York
  - New York Oncology Hematology P.C., Albany, New York
  - Local Institution - 0090, Rochester, New York
  - University of Rochester Cancer Center, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Local Institution - 0021, Charlotte, North Carolina
  - Local Institution - 0039, Cincinnati, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Local Institution - 0051, Portland, Oregon
  - Providence Cancer Center/Earle A. Chiles Res. Inst., Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Local Institution - 0029, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Greenville Health System - Cancer Institute - Faris Road, Greenville, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Local Institution - 0037, Greenville, South Carolina
  - Local Institution - 0083, Dallas, Texas
  - UNC School of Medicine, Dallas, Texas
  - Intermountain Healthcare - LDS Hospital Blood and Marrow Transplant, Salt Lake City, Utah
  - Intermountain Healthcare - LDS Hospital, Salt Lake City, Utah
  - Local Institution - 0074, Salt Lake City, Utah
  - Northwest Medical Specialties, Tacoma, Washington
  - UNC School of Medicine, Tacoma, Washington
  - Local Institution - 0055, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Froedtert Hospital, Milwaukee, Wisconsin
  - UNC School of Medicine, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sehgal A, Hoda D, Riedell PA, Ghosh N, Hamadani M, Hildebrandt GC, Godwin JE, Reagan PM, Wagner-Johnston ND, Essell J, Nath R, Solomon SR, Champion R, Licitra E, Fanning S, Gupta NK, Chow VA, Yuan B, Yang Z, Ogasawara K, Thorpe J, Gordon LI. Lisocabtagene maraleucel for R/R LBCL in patients not intended for HSCT: final results of the phase 2 PILOT study. Blood Adv. 2025 Aug 12;9(15):3694-3705. doi: 10.1182/bloodadvances.2024015262. PMID 40305658
- [Derived] Ghosh N, Sehgal A, Liu FF, Kostic A, Crotta A, De Benedetti M, Faccone J, Peng L, Gordon LI. Comparative efficacy of lisocabtagene maraleucel in the PILOT study versus second-line chemotherapy regimens in the real world. Haematologica. 2025 Mar 1;110(3):693-705. doi: 10.3324/haematol.2024.285828. PMID 39479862
- [Derived] Gordon LI, Liu FF, Braverman J, Hoda D, Ghosh N, Hamadani M, Hildebrandt GC, Peng L, Guo S, Shi L, Sehgal A. Lisocabtagene maraleucel for second-line relapsed or refractory large B-cell lymphoma: patient-reported outcomes from the PILOT study. Haematologica. 2024 Mar 1;109(3):857-866. doi: 10.3324/haematol.2023.283162. PMID 37646670
- [Derived] Sehgal A, Hoda D, Riedell PA, Ghosh N, Hamadani M, Hildebrandt GC, Godwin JE, Reagan PM, Wagner-Johnston N, Essell J, Nath R, Solomon SR, Champion R, Licitra E, Fanning S, Gupta N, Dubowy R, D'Andrea A, Wang L, Ogasawara K, Thorpe J, Gordon LI. Lisocabtagene maraleucel as second-line therapy in adults with relapsed or refractory large B-cell lymphoma who were not intended for haematopoietic stem cell transplantation (PILOT): an open-label, phase 2 study. Lancet Oncol. 2022 Aug;23(8):1066-1077. doi: 10.1016/S1470-2045(22)00339-4. Epub 2022 Jul 12. PMID 35839786
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All efficacy and safety analyses were conducted on the JCAR017-treated Analysis Set.
Groups:
- Lisocabtagene Maraleucel (JCAR017): Participants underwent leukapheresis and may receive salvage low- dose chemotherapy or one cycle of non-curative standard of care antitumor therapy if required. Eligible participants then received lymphodepleting chemotherapy with fludarabine and cyclophosphamide (flu/cy) followed by a single dose of JCAR017 (100×10^6 CAR+ T cells) administered intravenously (IV) 2 to 7 days after completion of lymphodepleting chemotherapy.
Period: Pre-Treatment Phase
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Started (Participants who underwent leukapheresis) | 74
Completed (Participants who completed leukapheresis and continued to lymphodepleting chemotherapy (LDC) treatment period) | 63
Not Completed | 11
Not completed — Other reasons | 1
Not completed — No longer meets eligibility criteria | 4
Not completed — Disease-related complications | 1
Not completed — Death | 5
Period: Treatment Phase
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Started (Participants who underwent lymphodepleting chemotherapy (LDC) treatment) | 63
Received JCAR017 | 61
Received Nonconforming Product | 1
Did Not Receive Either JAR017 or Nonconforming Product | 1
Completed (Completed study) | 30
Not Completed | 33
Not completed — Withdrawal by Subject | 7
Not completed — Other reasons | 1
Not completed — Death | 23
Not completed — Did not receive either JAR017 or nonconforming product | 1
Not completed — Received nonconforming product | 1

BASELINE CHARACTERISTICS:
Population: 74 participants were leukapheresed.
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (6.57)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 8
  >= 65 to < 70 years | 7
  >= 70 to < 75 years | 27
  >= 75 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 64
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is the percent of participants with a best overall response (BOR) of either complete response (CR) or partial reasons (PR) based on the Independent Review Committee (IRC) assessment recorded from the time of JCAR017 treatment until disease progression, end of study, the start of another anticancer therapy or JCAR017 retreatment.
  CR = Score 1, 2, or 3 with or without a residual mass on the positron emission tomography 5-point scale (PET 5PS). A score of 3 in many patients indicates a good prognosis with standard treatment.
  PR = Score 4 or 5b with reduced uptake compared with baseline and residual mass(es) of any size.
  PET 5PS = 1- no uptake above background; 2- uptake ≤ mediastinum; 3- uptake > mediastinum but ≤ liver; 4- uptake moderately > liver; 5- uptake markedly higher than liver and/or new lesions; X- new areas of uptake unlikely to be related to lymphoma.
Time Frame: From first dose to disease progression, end of study, the start of another anticancer therapy, or hematopoietic stem cell transplantation (up to approximately 24 months)
Population: All participants with PET positive disease who received at least one infusion of JCAR017
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 61
Percent of Participants | 80.3 [68.2 to 89.4]
Statistical Analysis 1: Comparison: Lisocabtagene Maraleucel (JCAR017); Test type: Superiority; p < .0001, Exact binomial test — One sided P-value is calculated based on the null hypothesis ORR <= 50.2%

2. Secondary Outcome: Number of Participants With Any Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event that started any time from initiation of product administration through and including 90 days following product administration. AEs that occurred after the initiation of subsequent anticancer therapy or product retreatment were not considered as product TEAE. AEs are graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (Version 4.03) (NCI CTCAE) guidelines where Grade 3= Severe, Grade 4= Life-threatening, and 5 = Death.
Time Frame: From first dose to 90 days following first dose (up to approximately 90 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 61
Participants
  Participants with any TEAE | 59
  Participants with any serious TEAEs | 20
  Participants with any Grade ≥ 3 TEAEs | 48
  Participants with any product-related TEAE | 48

3. Secondary Outcome: Change From Baseline of Hematology Laboratory Results: Hemoglobin
Description: Change from baseline in Hematology laboratory analysis. Includes Hemoglobin. Baseline is the last observation collected prior to or on the date of product infusion.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion evaluable for hematology laboratory tests
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 59
g/L | 1.9 (10.05)

4. Secondary Outcome: Change From Baseline of Hematology Laboratory Results: Leukocytes, Lymphocytes, Neutrophils, Platelets
Description: Change from baseline in Hematology laboratory analysis. Includes Leukocytes, Lymphocytes, Neutrophils, and Platelets. Baseline is the last observation collected prior to or on the date of product infusion.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion evaluable for hematology laboratory tests
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 59
10^9 cells/L
  Leukocytes | 0.921 (3.8562)
  Lymphocytes | 0.537 (0.5953)
  Neutrophils | -0.216 (3.4010)
  Platelets | -61.6 (96.55)

5. Secondary Outcome: Change From Baseline of Chemistry Laboratory Results: Albumin
Description: Change from baseline in Chemistry laboratory analysis. Includes Albumin. Baseline is the last observation collected prior to or on the date of product infusion.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion evaluable for chemistry laboratory tests
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 59
g/L | 3.05 (3.866)

6. Secondary Outcome: Change From Baseline of Chemistry Laboratory Results: Alanine Aminotransferase, Aspartate Aminotransferase, Lactate Dehydrogenase
Description: Change from baseline in Chemistry laboratory analysis. Includes Alanine Aminotransferase, Aspartate Aminotransferase, and Lactate Dehydrogenase. Baseline is the last observation collected prior to or on the date of product infusion.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion evaluable for chemistry laboratory tests
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 59
U/L
  Alanine Aminotransferase | 4.6 (16.42)
  Aspartate Aminotransferase | -3.9 (21.22)
  Lactate Dehydrogenase | -138.2 (339.82)

7. Secondary Outcome: Change From Baseline of Chemistry Laboratory Results: Bilirubin, Creatinine, Direct Bilirubin, Urate
Description: Change from baseline in Chemistry laboratory analysis. Includes Bilirubin, Creatinine, Direct Bilirubin, and Urate. Baseline is the last observation collected prior to or on the date of product infusion.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion evaluable for chemistry laboratory tests
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 59
umol/L
  Bilirubin | -0.1741 (6.36075)
  Creatinine | 5.8734 (21.32985)
  Direct Bilirubin: number analyzed (Participants) | 55
  Direct Bilirubin | 0.0306 (2.35650)
  Urate: number analyzed (Participants) | 56
  Urate | 5.7897 (93.90174)

8. Secondary Outcome: Change From Baseline of Chemistry Laboratory Results: Calcium Corrected, Magnesium, Phosphate, Potassium, Sodium
Description: Change from baseline in Chemistry laboratory analysis. Includes Calcium Corrected, Magnesium, Phosphate, Potassium, and Sodium. Baseline is the last observation collected prior to or on the date of product infusion.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion evaluable for chemistry laboratory tests
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 59
mmol/L
  Calcium Corrected | -0.0261 (0.12183)
  Magnesium: number analyzed (Participants) | 57
  Magnesium | -0.0209 (0.09292)
  Phosphate: number analyzed (Participants) | 58
  Phosphate | 0.0479 (0.22624)
  Potassium | -0.05 (0.426)
  Sodium | 1.0 (3.37)

9. Secondary Outcome: Complete Response (CR) Rate
Description: Complete response rate (CRR) was defined as the percent of participants with a best overall response (BOR) of complete response (CR) based on the Independent Review Committee (IRC) assessment recorded from the time of JCAR017 treatment until disease progression, end of study, the start of another anticancer therapy or JCAR017 retreatment.
  CR = Score 1, 2, or 3 with or without a residual mass on the positron emission tomography 5-point scale (PET 5PS). A score of 3 in many patients indicates a good prognosis with standard treatment.
  PET 5PS = 1- no uptake above background; 2- uptake ≤ mediastinum; 3- uptake > mediastinum but ≤ liver; 4- uptake moderately > liver; 5- uptake markedly higher than liver and/or new lesions; X- new areas of uptake unlikely to be related to lymphoma.
Time Frame: From first dose to disease progression, end of study, the start of another anticancer therapy, or hematopoietic stem cell transplant (up to approximately 24 months)
Population: All participants with PET positive disease who received at least one infusion of JCAR017
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 61
Percent of Participants | 54.1 [40.8 to 66.9]

10. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time from first complete response(CR) or partial response (PR) to progressive disease (PD) or death, whichever occurred first.
  CR = Score 1, 2, or 3 on the positron emission tomography 5-point scale (PET 5PS). A score of 3 indicates a good prognosis with standard treatment.
  PR = Score 4 or 5b with reduced uptake compared with baseline and residual mass(es) of any size.
  PD = Score 4 or 5b on PET 5PS with an increase in intensity of uptake from baseline and/or new fluorodeoxyglucose-avid foci consistent with lymphoma at interim or end-of-treatment assessment.
  PET 5PS = 1-no uptake above background; 2-uptake ≤ mediastinum; 3-uptake > mediastinum but ≤ liver; 4-uptake moderately > liver; 5-uptake markedly higher than liver and/or new lesions; X- new areas of uptake unlikely to be related to lymphoma.
Time Frame: From first dose to up to approximately 24 months
Population: All participants with PET positive disease who received at least one infusion of JCAR017 and achieved a response (CR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 49
Months | 23.26 [6.24 to NA] — Insufficient number of participants with events.

11. Secondary Outcome: Duration of Response (DOR) in Participants With Complete Response (CR)
Description: DOR for participants with a best overall response of CR was defined as the time from documentation of first response (or CR) to progressive disease (PD) or death, whichever occurred first. The first documentation of CR/PR is the latest of all dates of required measurements to establish the response. The progression date is the earliest date of all assessments that led to a response assessment of PD.
  CR = Score 1, 2, or 3 on the positron emission tomography 5-point scale (PET 5PS). A score of 3 indicates a good prognosis with standard treatment.
  PD = Score 4 or 5b on PET 5PS with an increase in intensity of uptake from baseline and/or new fluorodeoxyglucose-avid foci consistent with lymphoma at interim or end-of-treatment assessment.
  PET 5PS = 1-no uptake above background; 2-uptake ≤ mediastinum; 3-uptake > mediastinum but ≤ liver; 4-uptake moderately > liver; 5-uptake markedly higher than liver and/or new lesions; X- new areas of uptake unlikely to be related to lymphoma.
Time Frame: From first dose to up to approximately 24 months
Population: All participants with PET positive disease who received at least one infusion of JCAR017 and achieved complete response (CR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 33
Months | NA [21.65 to NA] — Insufficient number of participants with events.

12. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from JCAR017 infusion to progressive disease (PD) or death. Kaplan-Meier (KM) methodology will be used to analyze PFS.
  PD = Score 4 or 5b on the positron emission tomography 5-point scale (PET 5PS) with an increase in intensity of uptake from baseline and/or new fluorodeoxyglucose-avid foci consistent with lymphoma at interim or end-of-treatment assessment.
  PET 5PS = 1- no uptake above background; 2- uptake ≤ mediastinum; 3- uptake > mediastinum but ≤ liver; 4- uptake moderately > liver; 5- uptake markedly higher than liver and/or new lesions; X- new areas of uptake unlikely to be related to lymphoma.
Time Frame: From first dose to progressive disease (PD) or death (up to approximately 24 months)
Population: All participants with PET positive disease who received at least one infusion of JCAR017
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 61
Months | 9.03 [4.17 to NA] — Insufficient number of participants with events.

13. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS is defined as the time from JCAR017 infusion to the earliest of the following events: death from any cause, progressive disease (PD), or starting a new anticancer therapy. Kaplan-Meier (KM) methodology will be used to analyze EFS.
  PD = Score 4 or 5b on PET 5PS with an increase in intensity of uptake from baseline and/or new fluorodeoxyglucose-avid foci consistent with lymphoma at interim or end-of-treatment assessment.
  PET 5PS = 1-no uptake above background; 2-uptake ≤ mediastinum; 3-uptake > mediastinum but ≤ liver; 4-uptake moderately > liver; 5-uptake markedly higher than liver and/or new lesions; X- new areas of uptake unlikely to be related to lymphoma.
Time Frame: From first dose to death from any cause, progressive disease (PD), or starting a new anticancer therapy (up to approximately 24 months)
Population: All participants with PET positive disease who received at least one infusion of JCAR017
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 61
Months | 7.23 [3.22 to 24.28]

14. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from JCAR017 infusion to the date of death. Kaplan-Meier (KM) methodology will be used to analyze OS.
Time Frame: From first dose to date of death (up to approximately 24 months)
Population: All participants with PET positive disease who received at least one infusion of JCAR017
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 61
Months | NA [16.33 to NA] — Insufficient number of participants with events.

15. Secondary Outcome: PK Parameters of JCAR017 in Blood as Assessed by qPCR: Cmax
Description: Pharmacokinetic (PK) analyses were based on quantitative polymerase chain reaction (qPCR).
  Cmax = Maximum observed blood concentration.
Time Frame: From first dose to up to 24 months
Population: All participants who received at least one infusion of JCAR017 who have baseline and on-study PK measurements assessed by qPCR
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/μg
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 55
copies/μg | 22516.3 (237.4)

16. Secondary Outcome: PK Parameters of JCAR017 in Blood as Assessed by qPCR: Tmax
Description: Pharmacokinetic (PK) analyses were based on quantitative polymerase chain reaction (qPCR). Tmax = Time of maximum observed blood concentration.
Time Frame: From first dose to up to 24 months
Population: as for outcome 15
Measure: Median (Full Range); unit: Day
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 55
Day | 10.0 [6 to 22]

17. Secondary Outcome: PK Parameters of JCAR017 in Blood as Assessed by qPCR: AUC (0-28)
Description: Pharmacokinetic (PK) analyses were based on quantitative polymerase chain reaction (qPCR). AUC (0-28) = Area under the curve for concentration.
Time Frame: From first dose to up to 24 months
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*copies/ug
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 55
day*copies/ug | 178631.0 (228.3)

18. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Fatigue Subscale
Description: * Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire.
  * The EORTC QLQ-C30 is a 30-item scale composed of both multi-item scales and single-item measures.
  * All of the scales and single-item measures range in score from 0 to 100. A 10-point change in the scoring is considered to be a meaningful change in HRQoL.
  * Symptom scale/item higher score represents a high level of symptomatic problem.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion who has an analyzable baseline scale and at least one post-baseline analyzable scale
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 36.706 (27.6193)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 37.731 (19.9473)

19. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Physical Functioning Subscale
Description: * Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire.
  * The EORTC QLQ-C30 is a 30-item scale composed of both multi-item scales and single-item measures.
  * All of the scales and single-item measures range in score from 0 to 100. A 10-point change in the scoring is considered to be a meaningful change in HRQoL.
  * Functional scale and global health status/HRQoL higher scale score represents a higher level of well-being and better ability of daily functioning.
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 77.827 (24.2897)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 71.667 (23.8395)

20. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Cognitive Functioning Subscale
Description: as for outcome 19
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 83.333 (17.4078)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 88.194 (14.9698)

21. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Global Health/QoL Subscale
Description: as for outcome 19
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 66.815 (25.5491)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 72.049 (18.7910)

22. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Role Functioning Subscale
Description: as for outcome 19
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 77.083 (30.4117)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 69.792 (28.0695)

23. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Emotional Functioning Subscale
Description: as for outcome 19
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline: number analyzed (Participants) | 55
  Baseline | 81.061 (17.1575)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 86.806 (13.4077)

24. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Social Functioning Subscale
Description: as for outcome 19
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 74.702 (26.3985)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 72.917 (25.8713)

25. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Pain Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 26.488 (29.2631)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 13.542 (22.4546)

26. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Nausea/Vomiting Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 5.655 (10.6727)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 6.250 (14.4338)

27. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Constipation Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 11.905 (23.2931)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 6.944 (13.6805)

28. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Diarrhea Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 13.690 (21.8135)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 11.806 (21.1821)

29. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Insomnia Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 25.595 (27.7005)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 20.139 (27.2798)

30. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Dyspnea Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 10.714 (21.1843)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 13.194 (17.8510)

31. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Appetite Loss Subscale
Description: as for outcome 18
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline: number analyzed (Participants) | 55
  Baseline | 18.788 (29.9270)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 22.222 (28.6277)

32. Secondary Outcome: Mean Score in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Financial Difficulties Subscale
Description: as for outcome 19
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 56
Scores on a scale
  Baseline | 13.690 (22.7208)
  Day 29: number analyzed (Participants) | 48
  Day 29 | 14.583 (21.6421)

33. Secondary Outcome: Health-Related Quality of Life (HRQoL) Assessed by the FACT-Lym Subscale
Description: The Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym) consists of the FACT-General scale and a 15-item lymphoma-specific additional concerns subscale (LYM). This scale addresses symptoms and functional limitations that are important to lymphoma patients. The LYM items are scored on a 0 ("Not at all") to 4 ("Very much") response scale. Items are aggregated to a single score on a 0-60 scale.
Time Frame: Baseline and Day 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 49
Scores on a scale
  Baseline | 44.22 (8.804)
  Day 29: number analyzed (Participants) | 42
  Day 29 | 48.71 (6.447)

34. Secondary Outcome: Health-Related Quality of Life (HRQoL) Assessed by the EuroQol Instrument EQ-5D-5L
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. These health states are converted to a single index value using the crosswalk method to the EQ-5D-3L value set from the United Kingdom (UK). The EQ-5D-5L health states ranged from -.594 for the worst (55555) to 1 for the best (11111) for UK value set with an optimal health state is assigned a score of 1.00, death is assigned a score of 0.00 and negative values representing values as worse than dead. A change of .08 is considered to be a clinically meaningful change in health utility.
Time Frame: Baseline and Day 29
Population: All participants who received at least one JCAR017 infusion who completed 5-dimension measures at baseline and at least one post-baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 55
Scores on a scale
  Baseline | 0.7378 (0.23190)
  Day 29: number analyzed (Participants) | 46
  Day 29 | 0.7719 (0.20651)

35. Secondary Outcome: Numbers of Intensive Care Unit (ICU) Inpatient Days
Description: The numbers of ICU inpatient days.
Time Frame: From first dose after JCAR017 infusion to up to approximately 24 months
Population: All participants who received at least one infusion of JCAR017 who were monitored inpatient
Measure: Median (Full Range); unit: Day
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 41
Day | 0.0 [0 to 30]

36. Secondary Outcome: Numbers of Non-intensive Care Unit (ICU) Inpatient Days
Description: Number of non-ICU inpatient days.
Time Frame: From first dose after JCAR017 infusion to up to approximately 24 months
Population: All participants who received at least one infusion of JCAR017 who were monitored inpatient
Measure: Median (Full Range); unit: Day
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 41
Day | 14.0 [3 to 34]

37. Secondary Outcome: The Number of Participants That Were Hospitalized For Adverse Events, Prophylaxis, Other
Description: Length of hospitalization stay was reported for up to 24 months post liso-cel infusion. Reasons for hospitalization include adverse events, prophylaxis, and other. Adverse events were reported for up to 90 days post liso-cel infusion.
Time Frame: From first dose after JCAR017 infusion to up to approximately 24 months
Population: All participants who received at least one infusion of JCAR017 who were monitored inpatient
Measure: Number; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 41
Participants
  Adverse Event | 2
  Prophylaxis for CAR T-cell administration | 36
  Other | 3

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from the first participant undergoing leukapheresis until study completion (up to approximately 52 months). SAEs and Other AEs were assessed from the first participant undergoing leukapheresis to 90 days following the first participant undergoing leukapheresis (up to approximately 90 days).
Description: The total number at risk for all-cause mortality represents all participants who underwent leukapheresis. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants that received at least 1 dose of study medication (JCAR017).
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
All-Cause Mortality (participants affected / at risk) | 30/74
Serious Adverse Events (participants affected / at risk) | 20/61
Other Adverse Events (participants affected / at risk) | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lisocabtagene Maraleucel (JCAR017) (N=61)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Cytokine release syndrome (Immune system disorders) | 8
Bacteraemia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Stenotrophomonas sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lisocabtagene Maraleucel (JCAR017) (N=61)
Anaemia (Blood and lymphatic system disorders) | 19
Leukopenia (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 5
Fatigue (General disorders) | 24
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 5
Cytokine release syndrome (Immune system disorders) | 15
Hypogammaglobulinaemia (Immune system disorders) | 5
Fall (Injury, poisoning and procedural complications) | 5
Neutrophil count decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 10
Anxiety (Psychiatric disorders) | 5
Confusional state (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 10
Orthostatic hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT03483103/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT03483103/SAP_001.pdf